CLINICAL TRIAL: NCT00437164
Title: A Randomized, Double-blind, Parallel, Placebo-Controlled, Study to Evaluate the Safety and Tolerability of Oral GW677954 Capsules (15 mg) in Combination With Insulin in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study To Assess GW677954 Used In Combination With Insulin In Subjects Who Have Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision not related to safety.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADG106149
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-05

CONDITIONS: Type 2 Diabetes Mellitus; Diabetes Mellitus, Type 2
Keywords: NaBr; Sodium Bromide; DEXA Deuterium; Total Body Water; Insulin; D2O; GW677954; Randomized Withdrawal; T2DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Insulin
Drug: Oral GW677954 Capsules (15 mg)
  Other Names: Insulin

SUMMARY:
Many drugs used for the treatment of Type 2 Diabetes Mellitus cause the body to retain water. This study will assess whether or not GW677954 causes the body to retain fluid.

ELIGIBILITY:
Inclusion criteria:

* Have been diagnosed by a doctor with Type 2 Diabetes Mellitus at least 3 months before Screening
* Have a body mass index within range 25 to 40.0kg/m2 inclusive
* Females who meet above criteria must be physiologically incapable of becoming pregnant (ie., surgically sterilized, or post-menopausal per protocol definition)

Exclusion criteria:

* Significant weight loss or gain in the 3 months before screening
* Have used insulin to treat hyperglycemia within 3 months before screening
* Have a history of fluid retention
* Have uncontrolled high blood pressure
* Have liver disease
* Take loop diuretics (water pills), certain blood thinners, and/or St. Johns Wort. - Have or have had certain kinds of cancer

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2006-09; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
changes in fluid related parameters as measured by hematocrit and hemoglobin levels and body weight | up to 24 weeks

SECONDARY OUTCOMES:
safety/tolerability, as measured by adverse events, clinical laboratory, edema & glycemic measures, ophthalmic assessments; & changes in weight, waist & hip circumference | up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Beverly Hills, California, United States